CLINICAL TRIAL: NCT01314963
Title: Efficacy of a Novel, High-Sensitivity, Portable, Hand-Held Gamma Camera Used Intraoperatively for Identification of Sentinel Lymph Nodes With Lymphoscintigraphy
Brief Title: Efficacy of Gamma Camera Used Intraoperatively for ID of Sentinel Lymph Nodes w/ Lymphoscintigraphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Whitaker Foundation (Unknown)
Responsible Party: Principal Investigator, John B. Sunwoo, Assistant Professor of Otolaryngology - Head and Neck Surgery, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-06037; SU-03092011-7560 (Other: Stanford University); MEL0004 (Other: OnCore)
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma; Breast Cancer
MeSH Terms: conditions — Multiple Myeloma; Breast Neoplasms | interventions — Lymphoscintigraphy

STUDY DESIGN:
Intervention Model Description: The unit of study in this trial was sentinel lymph nodes (SLNs) rather individual participants. with the comparison conducted by evaluation of each SLN with the prototype intraoperative handheld gamma camera (pIHGC) and standard of care intraoperative gamma probes (GP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intraoperative handheld Gamma Camera (pIHGC) (Experimental): The prototype intraoperative handheld gamma camera (pIHGC)
  Interventions: Device: Prototype intraoperative handheld gamma camera (pIHGC); Radiation: radioactive Tc99M
- Gamma probes (GP) (Active Comparator): Standard of care intraoperative gamma probes (GP) currently in use.
  Interventions: Device: Lymphoscintigraphy with intraoperative gamma probes (GP); Radiation: radioactive Tc99M

INTERVENTIONS:
Device: Prototype intraoperative handheld gamma camera (pIHGC) — The prototype intraoperative handheld gamma camera (pIHGC) consists of a parallel-hole lead collimator coupled to a pixilated sodium iodide-thallium [NaI(Tl)] scintillation crystal array, itself coupled to a flat panel, multi-anode Hamamatsu H8500 position-sensitive photomultiplier tube. The collimator is 5x5 cm2 large in area and 1.5 cm thick, with 1.3 mm hexagonal holes and 0.2 mm septa. The 1.7 mm pitch crystal array is composed of 29x29 individual crystals, each 1.5x1.5x6 mm3 in size.
  Arms: Intraoperative handheld Gamma Camera (pIHGC)
Device: Lymphoscintigraphy with intraoperative gamma probes (GP) — Lymphoscintigraphy with standard of care intraoperative gamma probes (GP)
  Arms: Gamma probes (GP)
Radiation: radioactive Tc99M — Lymphoscintigraphy involves injection of 0.4 to 1.0 mCi of radioactive Tc99M sulfur colloid around at the tumor site.

SUMMARY:
This study evaluates the ability of a prototype intraoperative handheld gamma camera (pIHGC) to image (detect) sentinel lymph nodes (SLNs) in melanoma and breast cancer during surgical excision, as compared to standard of care intraoperative gamma probes (GP). The unit of study in this trial was SNLs rather individual participants. Each device was assessed for relative node detection sensitivity (S) of those SLNs.

DETAILED DESCRIPTION:
Lymphoscintigraphy is an accepted and commonly-performed procedure used for staging of certain cancers, especially melanoma and breast cancer. It involves injecting a small amount of radioactivity under the skin in order to identify lymph nodes which should be biopsied (ie, the "sentinel lymph node, SLN") to determine if cancer has spread. The study objective was to evaluate the potential benefit of a new, camera-based technology (prototype device) which allows actual images to be obtained intra-operatively in the identification of sentinel nodes.

Each device was assessed for relative node detection sensitivity (S), defined as the proportion of sentinel lymph nodes (SLNs) that were identified with each instrument, with the proportion determined as the number of true positives (TP) divided by the total evaluated (N).

ELIGIBILITY:
INCLUSION CRITERIA

* Malignancy for which sentinel node biopsy with lymphoscintigraphy are indicated as part of the standard of care for tumor staging
* Age 18 or greater.
* Healthy enough for surgery
* Able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA

* No exclusion requirements due to co-morbid disease or intercurrent illness.
* Documented allergy to colloid.
* Lymphoscintigraphy presents excessive high risk, eg, a consideration if pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-07-26 (Actual); Study Completion 2012-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Sunwoo, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Olcott P, Pratx G, Johnson D, Mittra E, Niederkohr R, Levin CS. Clinical evaluation of a novel intraoperative handheld gamma camera for sentinel lymph node biopsy. Phys Med. 2014 May;30(3):340-5. doi: 10.1016/j.ejmp.2013.10.005. Epub 2013 Nov 14. PMID 24239343

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This study evaluates the ability of 2 procedures to detect sentinel lymph nodes (SLNs), and does not evaluate between groups of participants.
Period: Overall Study
Arm/Group | All Participants
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The required data for baseline results is participant-level data. This study is a comparison of lesion-level data sets, ie, a comparison of intra-participant data. It is not possible to segregate participant baseline data to one group or the other of the intra-participant datasets.
Arm/Group | All Participants
Number analyzed (Participants) | 50
Age, Customized [Count of Participants; unit: Participants] — All available information on age is provided. Some data are missing, specifically whether or not certain participants were older or younger than age 65. Therefore the number of participants 18 to 65 vs the number of participants older than 65 is not available.
  Participants
    18 years old or greater | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Relative Node Detection Sensitivity
Description: Relative node detection sensitivity (S) was defined as the proportion of sentinel lymph nodes (SLNs) that were identified with each instrument, with the proportion determined as the number of true positives (TP) divided by the total evaluated (N). The outcome result is expressed as the percentage for each device with 95% confidence intervals.
Time Frame: 1 day
Population: Sentinel lymph nodes (SLNs) were evaluated for detection by the 2 methods.
Measure: Number (95% Confidence Interval); unit: Percentage (%) of SLNs detected
Units Other Than Participants: Sentinel lymph nodes (SLNs)
Groups:
- Gamma Probes (GP): Lymphoscintigraphy with standard of care intraoperative gamma probes (GP)
  radioactive Tc99M: Lymphoscintigraphy involves injection of 0.4 to 1.0 mCi of radioactive Tc99M sulfur colloid around at the tumor site.
Arm/Group | Intraoperative Handheld Gamma Camera (pIHGC) | Gamma Probes (GP)
Number analyzed (Participants) | 50 | 50
Number analyzed (Sentinel lymph nodes (SLNs)) | 104 | 104
Percentage (%) of SLNs detected | 88.5 [82.3 to 94.6] | 94.2 [89.7 to 98.7]

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- All Participants - Intraoperative Handheld Gamma Camera (pIHGC: The entire set of sentinel lymph nodes (SLNs) excised from study participants (ie, all participants) were evaluated with the intraoperative handheld gamma camera (pIHGC).
- All Participants - Gamma Probes (GP): The entire set of sentinel lymph nodes (SLNs) excised from study participants (ie, all participants) were evaluated with the gamma probes (GP).
Arm/Group | All Participants - Intraoperative Handheld Gamma Camera (pIHGC | All Participants - Gamma Probes (GP)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No